CLINICAL TRIAL: NCT06869629
Title: SENOMAC-ULTRA: A Prospective Randomised Trial on the Omission of Axillary Lymph Node Dissection in Ultrasound-detectable Axillary Metastases in Primary Breast Cancer Treated by Upfront Surgery
Brief Title: Omission of Axillary Lymph Node Dissection in Case of Tumor Spread to Lymph Nodes in the Armpit in Breast Cancer
Acronym: SENOMAC-ULTRA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jana de Boniface, Professor, MD, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SENOMAC-ULTRA
Record Dates: First submitted 2025-03-04; First posted 2025-03-11 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Breast Carcinoma; Breast Cancer; Breast Surgery
Keywords: axillary metastases; axillary lymph node dissection; targeted axillary dissection; sentinel lymph node biopsy; axillary ultrasonography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Non-inferiority open randomised design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Axillary lymph node dissection (Active Comparator): Axillary lymph node dissection
  Interventions: Procedure: Axillary lymph node dissection
- Targeted axillary dissection (Experimental): Removal of the marked metastasis/-es and a sentinel lymph node biopsy
  Interventions: Procedure: Targeted axillary dissection

INTERVENTIONS:
Procedure: Targeted axillary dissection — Known metastases are marked before surgery and removed together with a sentinel lymph node biopsy
  Arms: Targeted axillary dissection
Procedure: Axillary lymph node dissection — Routine axillary clearance removing about 10+ lymph nodes from axillary levels I and II
  Arms: Axillary lymph node dissection

SUMMARY:
SENOMAC-ULTRA enrols patients who are planned for upfront surgery for a breast cancer that has spread to lymph nodes in the armpit, and that have been detected already prior to surgery by imaging, e.g. ultrasonography. In this situation, a full axillary lymph node dissection, removing more than 10 lymph nodes from the arm pit, is unnecessarily extensive in about half of the patients. More extensive surgery leads to a risk for arm lymphedema and functional problems with the arm and shoulder region, which should be avoided if not beneficial for diagnosis or prognosis. This trial seeks to ascertain that less extensive surgery, performed by only removing the first lymph node/s in the armpit (the sentinel lymph node/s) and the known metastatic lymph nodes (targeted axillary dissection, TAD), offers non-inferior survival outcomes to a full axillary lymph node dissection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary invasive breast cancer clinical stage II-III
* Palpable or non-palpable axillary metastases visible by ultrasound (other imaging accepted if confirmatory ultrasound is performed) and confirmed by fine needle aspiration or core biopsy
* Written informed consent
* Age ≥ 18 years

Exclusion Criteria:

* Distant metastases
* Ipsilateral metastases in internal mammary, infra- or supraclavicular lymph nodes without confirmed axillary nodal involvement
* Preoperative suspicion of extensive nodal involvement, i.e. locally advanced disease
* Nodes fixed to each other or to neighbouring structures on palpation or imaging
* History of contralateral invasive breast cancer within 5 years
* Bilateral invasive breast cancer if (i) one side meets any exclusion criteria or (ii) both sides meet all inclusion criteria
* Pregnancy
* Neoadjuvant systemic treatment (short course of neoadjuvant endocrine therapy <three months is allowed)
* Medical contraindications for or expressed preoperative wish to abstain from radiotherapy or the recommended adjuvant systemic treatment which complies with standard of care, taking age and comorbidity into consideration
* Inability to absorb or understand the meaning of the study information; for example, through disability, inadequate language skills or dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1380 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | 5 years
  Time to event where an event is death if any cause or a recurrence of breast cancer

SECONDARY OUTCOMES:
Arm morbidity | 1, 3, 5 years
  Arm function as reported by patients via the Lymphedema Functioning, Disability and Health questionnaire (Lymph-ICF), which consists of 29 questions about impairments in function, activity limitations, and participation restrictions of patients with breast cancer and arm lymphedema. The questionnaire is divided into 5 domains: physical function, mental function, household activities, mobility activities, and life and social activities. Each item is scored on a visual analogue scale (0-100 mm) resulting in domain scores ranging from 0 to 100. Higher scores indicate more severe arm dysfunction. Lymph-ICF scores also categorize into "no problem", "a small problem", "a moderate problem", "a severe problem", and "a very severe problem".
Health-related quality of life | 1, 3, 5 years
  Health-related quality of life measured by EORTC C30. The EORTC QLQ-C30 questionnaire measures HRQoL among cancer patients in general and consists of 30 items divided into multi-item scales and single items. The multi-item scales include one global health and quality of life (QoL) scale, five function subscales (physical, role, emotional, cognitive, social) and three symptom subscales (fatigue, nausea and vomiting, pain). The single items are dyspnoea, insomnia, appetite loss, constipation, diarrhoea, financial difficulties. Each scale produces a total score from 0 to 100. High scores on functional subscales indicate better function, and high scores on symptom subscales indicate more severe problems.
Overall survival | 5 years
  Time to event where an event is death of any cause
Health-related quality of life - breast cancer | 1, 3, 5 years
  The EORTC QLQ-BR23 questionnaire measures functions and symptoms related to breast cancer treatment and consists of 23 items divided into two functional subscales (body image and sexuality) and three symptom subscales (systemic therapy side effects, arm symptoms, breast symptoms) and three single items (sexual enjoyment, upset by hair loss, future perspective). The functional and symptom subscales as well as the single items correspond to a response scale 1-4 (not at all, a little, quite a bit, very much). Each scale produces a total score from 0 to 100. High scores on functional subscales indicate better function, and high scores on symptom subscales indicate more severe problems.

CONTACTS AND LOCATIONS:
Overall Officials: Jana de Boniface, Principal Investigator — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: Yes
IPD may be shared upon reasonable request and with all relevnt legal and ethical requirements fulfilled. No request will be accepted before the publication of the primary endpoint.
Supporting Information: Study Protocol, SAP, ICF